CLINICAL TRIAL: NCT03905811
Title: A Pilot Study of Terazosin for Parkinson's Disease
Acronym: TZ-PD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jordan Schultz (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Jordan Schultz, PharmD, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201902772
Record Dates: First submitted 2019-04-01; First posted 2019-04-05 (Actual); Results first posted 2021-08-02 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease
Keywords: terazosin
MeSH Terms: conditions — Parkinson Disease | interventions — Terazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active (Experimental): Terazosin administered 5 mg once daily p.o. for 12 weeks
  Interventions: Drug: Terazosin 5 MG
- Placebo (Placebo Comparator): Placebo administered once daily p.o. for 12 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Terazosin 5 MG — 5 milligrams by mouth daily at bedtime
  Other Names: Hytrin
  Arms: Active
Drug: Placebo oral capsule — 1 capsule by mouth daily at bedtime
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The TZ-PD trial will be a 1:1 (active:placebo) randomized, double-blind, placebo-controlled Phase II trial to evaluate the safety and tolerability of terazosin for the treatment of PD.

DETAILED DESCRIPTION:
This will be a single center, randomized, double-blind, controlled, pilot study to assess the safety and tolerability of terazosin (TZ) at a dose of 5 milligrams (MG) daily for patients with PD. The primary goal of this study is to assess the safety and tolerability of TZ in patients with PD. This is a pilot study and is not powered to assess efficacy of this medication. Our hope is that this study will guide future studies of this (and similar) medications for the disease modification of PD. This study is also aimed to learn more about how patients with produce and use energy and if TZ can help to reverse energy deficits that appear in PD.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 40 and older with the diagnosis of idiopathic PD per UK Brain Bank criteria
* Hoehn-Yahr Stage I-III, on stable dopaminergic treatment regimen for ≥4 weeks prior to baseline.

Exclusion Criteria:

* Subjects unwilling or unable to give informed consent
* Secondary parkinsonism (e.g., drug induced)
* Parkinson-plus syndromes
* History of brain surgery for PD such as deep brain stimulation
* No confounding acute or unstable medical, psychiatric, orthopedic condition. Subjects who have hypertension, diabetes mellitus, depression, or other common age-related illness will be included if their disease under control with stable treatment regimen for at least 30 days.
* Neurogenic orthostatic hypotension defined as symptomatic decrease in BP > 20mmHg systolic or > 10mmHg diastolic and HR increase < 20bpm on supine to sitting or standing.
* Clinically significant traumatic brain injury or post-traumatic stress disorder
* Presence of other known medical or psychiatric comorbidity that in the investigator's opinion would compromise participation in the study
* Presence of dementia per Movement Disorder Society Level I criteria
* Major depression, bipolar affective disorder, or other mental health disorders that are sufficiently severe to increase adverse event risk or impact neuropathy assessment in the opinion of the responsible site principal investigator.
* Subjects with clinically significant depression as determined by a Beck Depression Inventory score greater than 21 at the screening visit
* Current suicidal ideation within one year prior to the baseline visit as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS)
* If the participant has a Beck Anxiety Score greater than 22 at the initial screening visit.
* History of exposure to typical or atypical antipsychotics or other dopamine blocking agents within 6 months prior to the baseline visit
* Use of investigational drugs within 30 days before screening
* Subjects have to be on a stable regimen of central nervous system acting medications (benzodiazepines, antidepressants, hypnotics) for 30 days prior to the baseline visit
* Use of doxazosin, alfuzosin, prazosin, or tamsulosin
* For female participant, pregnancy, or plans for child-bearing during study period
* Participant is restricted from traveling to and from the study site

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Schultz, PharmD, Principal Investigator — University of Iowa; Nandakumar Narayanan, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request with justification for request from qualified researchers, anonymized data will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after completion of this study
Access Criteria: Qualified researchers may contact the PI of this study with reasonable requests for data to be shared. Inquiries must include what hypothesis the researcher intends to test using the shared data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Placebo
Started | 8 | 5
Completed | 6 | 5
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (6.1) | 68.8 (6.6) | 66.4 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Intervention-related Adverse Events Between Treatment Arms
Description: All patient-reported adverse events will be determine to be related to the study intervention by the site investigator.
Time Frame: 12 weeks
Measure: Number; unit: Event
Arm/Group | Active | Placebo
Number analyzed (Participants) | 8 | 5
Event | 11 | 4

2. Primary Outcome: Incidence of Falls Between Treatment Arms
Description: The number of participants in each group who report a fall, as determined by the site investigator, will be reported.
Time Frame: 12 weeks
Measure: Number; unit: Event
Arm/Group | Active | Placebo
Number analyzed (Participants) | 8 | 5
Event | 0 | 0

3. Primary Outcome: Frequency of Drop-out From Study/Discontinuation of Study Intervention for Any Reason
Description: The number of participants in each group who drop out of the study for any reason will be compared.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 8 | 5
Participants | 3 | 0

4. Secondary Outcome: To Assess the Mean Change in Blood Pressure
Description: Mean change in sitting systolic blood pressure and diastolic blood pressure from baseline reading at 2 weeks, 6 weeks, and 12 weeks. A negative number indicates a decrease in blood pressure while a positive number indicates an increase in blood pressure.
Time Frame: At Baseline, 2 weeks, 6 weeks, and 12 weeks
Population: Change in Systolic BP at 2 weeks, 6 weeks, and 12 weeks Change in Diastolic BP at 2 weeks, 6 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Active | Placebo
Number analyzed (Participants) | 8 | 5
mmHg
  Systolic at 2 weeks | -5.29 (12.6) | -2.20 (11.5)
  Systolic at 6 weeks: number analyzed (Participants) | 7 | 5
  Systolic at 6 weeks | -15.05 (8.21) | 2.20 (23.2)
  Systolic at 12 weeks: number analyzed (Participants) | 5 | 5
  Systolic at 12 weeks | -11.0 (16.1) | -3.20 (13.1)
  Diastolic at 2 weeks | -2.00 (5.54) | -2.20 (8.87)
  Diastolic at 6 weeks: number analyzed (Participants) | 7 | 5
  Diastolic at 6 weeks | -5.29 (4.54) | 4.20 (8.14)
  Diastolic at 12 weeks: number analyzed (Participants) | 5 | 5
  Diastolic at 12 weeks | -9.40 (2.07) | -2.00 (11.3)

5. Secondary Outcome: Number of Participants With Intolerable Side Effects
Description: How many participants discontinued study as a result of intolerable adverse events that were deemed to be medication-related.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 8 | 5
Participants | 3 | 0

6. Secondary Outcome: Participants Demonstrating Non-Compliance
Description: All participants will be asked to bring their study intervention bottles to their 6 week visit and their 12 week visit so the Investigational Drug Pharmacy can count remaining pills and assess compliance based on dispensing history. A participant will be considered non-compliant if they had more than 5 missed doses during the course of the study.
Time Frame: At 2 weeks, 6 weeks and 12 weeks
Population: Number of participants analyzed changes at different time points due to participant drop-out
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 8 | 5
Participants
  Non-compliance at 2 weeks | 0 | 0
  Non-compliance at 6 weeks: number analyzed (Participants) | 7 | 5
  Non-compliance at 6 weeks | 0 | 0
  Non-compliance at 12 weeks: number analyzed (Participants) | 5 | 5
  Non-compliance at 12 weeks | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 week
Arm/Group | Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 8/8 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=8) | Placebo (N=5)
Dizzy/Lightheadedness (Nervous system disorders) | 7 | 1
Unsteady (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 1
Fatigue (Nervous system disorders) | 1 | 0
Orthostatic Hypotension (Nervous system disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
-Recruitment halted early due to the onset of the COVID-19 Pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT03905811/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03905811/ICF_002.pdf